CLINICAL TRIAL: NCT06047522
Title: Benefit of Virtual Reality Headset Use on Apathy in Older Adults With Major Neurocognitive Disorders
Acronym: APATHIE_RV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RIVAGES (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A02814-37
Record Dates: First submitted 2023-07-20; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Apathy in Dementia; Aged; Virtual Reality; Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The participant will benefit from three immersion sessions with the virtual reality headset, either individually or in a group session, accompanied by a team member trained in the use of the headset (psychomotrician, occupational therapist, doctor, psychologist, facilitator). At each session, the scale of observed emotions and the cybermalaise questionnaire will be completed (T1, T2, T3). At sessions 1 (T1) and 3 (T3), the investigator will administer the ECPAI behavior scale.
  Interventions: Device: Casque Lumeen

INTERVENTIONS:
Device: Casque Lumeen — Participants will take part in virtual reality sessions via headset. They will benefit from a before/after evaluation, and a 3-week intervention where they will have 1 virtual reality session per week.

SUMMARY:
The goal of this clinical trial is to verify that virtual reality is tolerably compatible with apathetic pathologies in patients and residents with major neurocognitive disorders. The main questions it aims to answer are:

* Does virtual reality have an impact on symptoms of apathy in the elderly?
* Is virtual reality well tolerated by the elderly? Participants will benefit from a 3-session virtual reality headset program with a healthcare professional. They will have one session per week for 3 weeks. They will be observed by another professional, who will complete observation grids on apathy, engagement in activity and tolerance of the virtual reality headset.

There is not a comparison group: Researchers will compare the scores before and after the intervention: the participant will be his own control.

DETAILED DESCRIPTION:
This study is a multicenter interventional exploratory study in two nursing homes and a geriatric long-term care service. Thirty patients will be included. They will be recruited from residents of the long-term care departments of two hospitals, and 4 nursing homes.

A pre- and post-intervention comparison will be made by assessing apathy using the apathy inventory and the neuropsychiatric inventory in the care team version. A comparison of participants' engagement will be carried out through ecological observation of the interventions. This will be objectivized by the Caregiver Interaction Behavior Scale (ECPAI) before the immersion program, and during the first and third virtual reality sessions. An ECPAI scale taken during a conventional animation prior to the program will establish a baseline state for the participant.

The main goal is to verify that virtual reality is tolerably compatible with apathetic pathologies in patients and residents with major neurocognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Persons over 65 years of age
* Persons living in nursing homes or hospitalized in long-term care
* Persons with correct vision or vision corrected by glasses
* People with no hearing problems, or with hearing loss corrected by a hearing aid
* Person with a major neurocognitive disorder
* Person with a Mini Mental State Examination (MMSE) cognitive score <26
* Individuals with documented apathy

Exclusion Criteria:

* Person with a history of epilepsy
* Persons wearing a pacemaker
* Person with open wounds of the face or skull
* Disabling headache or neck pain
* Person at the immediate end of life or in active palliative care
* Person with a contagious disease
* People who are bedridden or unable to get into a wheelchair
* Persons with severe neurological impairment
* Person with severe behavioral disorders endangering self or staff
* Persons unable to give oral consent

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Tolerance of virtual reality sessions | through study completion, an average of 6 months
  No change in Simulator Sickness Questionnaire (SSQ), or maintenance of "none" and "slight" scores. There are 16 items, each item is rated with the scale from none, slight, moderate to severe. After some calculations you have 3 subscores : Computation of nausea (N), oculomotor r disturbance (O), disorientation (D), and total simulator sickness (TS) scores.
Effectiveness of virtual reality sessions on apathy symptoms | through study completion, an average of 6 months
  Decrease in apathy scores on the Apathy Inventory (IA) (NPI). IA clinician assessment (0 to 4 score) has to take into account several factors: useful observation points, Patient history and social environment, personality, Information coming from the caregiver, Patient's responses to the clinical domains, autonomy.
  A score equal or upper to 4 is pathological.
Effectiveness of virtual reality sessions on apathy symptoms | through study completion, an average of 6 months
  Decrease in apathy scores on the Neuropsychiatric Inventory (NPI), caregiver version.
  The NPI-ES is based on responses from a member of the healthcare team involved in the patient's care. Responses refer to behaviours that have been present over the past week or other well-defined during other well-defined periods (e.g. 1 month ago, or since the last assessment). Answers should be brief, and can be formulated as "yes" or "no". In clinical practice, the most relevant factor to consider is the frequency x severity score for each area (a score greater than 2 is pathological).

SECONDARY OUTCOMES:
Security | through study completion, an average of 6 months
  no technical problems endangering the user during sessions, resulting in the session being stopped

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Maison de retraite la Passerelle, Larajasse, Rhône
  - Maison de retraite l'arc en ciel, Saint-Martin-en-Haut, Rhône
  - USLD Arcadie - CHU Rouen, Mont-Saint-Aignan, Seine Maritime
  - EHPAD d'Enghien, Enghien-les-Bains, Val d'Oise
  - EHPAD Louis Grassi, Presles, Val d'Oise
  - Hôpital Charles Foix, Ivry-sur-Seine, Val De Marne

IPD SHARING:
Plan to Share IPD: No
Each co-investigator coordinates his or her inclusions with the principal investigator, and sends him or her the data collected via secure messaging. The co-investigator is responsible for collating all the data.